CLINICAL TRIAL: NCT04832724
Title: A Phase 2, Open-label Study to Explore the Pharmacodynamics of Two Doses in Two Formulations of RGX-314 Gene Therapy Administered Via Subretinal Delivery in Participants With Neovascular Age-related Macular Degeneration
Brief Title: RGX-314 Gene Therapy Pharmacodynamic Study for Neovascular Age-related Macular Degeneration (nAMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RGX-314-2103
Record Dates: First submitted 2021-03-30; First posted 2021-04-06 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Neovascular Age-related Macular Degeneration; Wet Macular Degeneration; Wet Age-related Macular Degeneration
Keywords: AMD; wet AMD; wAMD; neovascular AMD; nAMD; gene therapy
MeSH Terms: conditions — Wet Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Commercial Formulation Dose 1 (Experimental): Dose 1 of RGX-314
  Interventions: Genetic: RGX-314
- Clinical Formulation Dose 1 (Experimental): Dose 1 of RGX-314
  Interventions: Genetic: RGX-314
- Commercial Formulation Dose 2 (Experimental): Dose 2 of RGX-314
  Interventions: Genetic: RGX-314
- Clinical Formulation Dose 2 (Experimental): Dose 2 of RGX-314
  Interventions: Genetic: RGX-314

INTERVENTIONS:
Genetic: RGX-314 — RGX-314 is a recombinant adeno-associated virus gene therapy vector carrying a coding sequence for a soluble anti-VEGF protein

SUMMARY:
RGX-314 is being developed as a novel one-time gene therapy for the treatment of neovascular (wet) age-related macular degeneration (nAMD) also referred to as Wet AMD. Wet AMD is characterized by loss of vision due to new, leaky blood vessel formation in the retina. The purpose of this phase 2, open label study is to evaluate whether different doses of RGX-314 from two different formulations (clinical versus eventual commercial formulation) perform the same in humans when delivered by subretinal administration

DETAILED DESCRIPTION:
Wet AMD is a significant cause of vision loss in the United States, Europe and Japan, with up to 2 million people living with wet AMD in these geographies alone. Current anti-VEGF therapies have significantly changed the landscape for treatment of wet AMD, becoming the standard of care due to their ability to prevent progression of vision loss in the majority of patients. These therapies, however, require life-long repeated intraocular injections to maintain efficacy. Due to the burden of treatment, patients often experience a decline in vision with reduced frequency of treatment over time. RGX-314 is being developed as a potential one-time treatment for wet AMD. RGX-314 uses an AAV8 vector that contains a gene that encodes for a monoclonal antibody fragment which binds to and neutralizes VEGF activity. This phase 2, open label study will explore the pharmacodynamics of two doses in two formulations of RGX-314 gene therapy via subretinal delivery in patients with neovascular Age-related Macular Degeneration. Approximately 60 patients (15 per cohort) who meet the inclusion/exclusion criteria will be enrolled in 4 sequential dose cohorts. A dose cohort will be comprised of 1 of 2 doses of RGX-314 in 1 of 2 formulations in order to explore the pharmacodynamics of RGX-314 based on aqueous humor transgene product (TP) concentrations. If the participants meet the study criteria and choose to participate in the study, their participation in the study will last about 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, aged ≥ 50 years and ≤ 89 years.
2. An Early Treatment Diabetic Retinopathy Study (ETDRS) BCVA-letter score between ≤ 78 and ≥ 40 in the study eye at Screening.
3. Diagnosis of choroidal neovascularization (CNV) secondary to age-related macular degeneration in the study eye previously treated with anti-VEGF.
4. Participants must have demonstrated a meaningful response to anti-VEGF therapy at study entry.
5. Willing and able to provide written, signed informed consent for this study.
6. Must be pseudophakic (at least 12 weeks postcataract surgery) in the study eye.

Exclusion Criteria:

1. CNV or macular edema in the study eye secondary to any causes other than AMD.
2. Subfoveal fibrosis or atrophy in study eye.
3. Any condition in the investigator's opinion that could limit visual acuity improvement in the study eye.
4. Active or history of retinal detachment or retinal tear in the study eye.
5. Advanced glaucoma in the study eye.
6. Prior treatment with gene therapy.
7. Myocardial infarction, cerebrovascular accident, or transient ischemic attack within the past 6 months.

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
RGX-314 target protein concentration in aqueous humor | At Week 24

SECONDARY OUTCOMES:
Incidence and severity of ocular Adverse Events (AEs) and overall AEs | Through Week 48
  Evaluate the safety and tolerability of RGX-314
Changes in Best Corrected Visual Acuity (BCVA) | At Week 24 and 48
  BCVA measured by Early Treatment Diabetic Retinopathy Study (ETDRS)
Changes in Central Retinal Thickness (CRT) | At Week 24 and 48
  CRT is measured by spectral domain optical coherence tomography (SD-OCT)
Mean Supplemental anti-VEGF injection annualized rate through week 24 and week 48 | Through Week 24 and week 48
  To assess the need for supplemental anti-VEGF therapy over 48 weeks

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - Barnet Dulaney Perkins Eye Center, Sun City, Arizona
  - Retina Consultants of San Diego, San Diego, California
  - California Retina Consultants, Santa Barbara, California
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Wilmer Eye Institute, Baltimore, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Sierra Eye Associates, Reno, Nevada
  - Eye Associates of New Mexico, Albuquerque, New Mexico
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Charles Retina Institute, Germantown, Tennessee
  - Texas Retina Associates, Dallas, Texas
  - Retina Consultants of Texas, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No